CLINICAL TRIAL: NCT05598957
Title: Evaluation of the Relationship of Vitamin D and Vitamin D Binding Protein with Disease Severity in Pediatric Sars-CoV2
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, mahmut caner us, Principal Investigator, Marmara University
Other Study IDs: 2022/10/17
Record Dates: First submitted 2022-10-06; First posted 2022-10-31 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2023-03

CONDITIONS: SARS CoV-2 Infection
Keywords: Sars Cov-2; Vitamin D Binding protein; free vitamin D; bioavailable vitamin D; children
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — to investigate the free and bioavailable vitamin D, 25OH vitamin d (μg/L), albumin (g/l) and VDBP levels, a 5 ml blood sample was collected from patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- uninfected Sars-CoV-2 group (Group 1): The study group was divided into three groups according to COVID-19 WHO clinical progression Scale: no viral RNA detected, uninfected Sars-CoV-2 patients (Group 1)
  Interventions: Diagnostic Test: Vitamin D Binding protein
- mild Sars-CoV-2 group (Group 2): The study group was divided into three groups according to COVID-19 WHO clinical progression Scale: viral RNA detected but asymptomatic disease, ambulatory mild disease (Group 2)
  Interventions: Diagnostic Test: Vitamin D Binding protein
- moderate to severe Sars-CoV-2 group (Group 3): The study group was divided into three groups according to COVID-19 WHO clinical progression Scale: hospitalized moderate disease, moderate to severe Sars-CoV-2 patients (group 3)
  Interventions: Diagnostic Test: Vitamin D Binding protein

INTERVENTIONS:
Diagnostic Test: Vitamin D Binding protein — Vitamin D-free and bioavailable metabolites were calculated by using Bikle and Vermeulen methods with using albumin, 25-OH vitamin D, vitamin D binding protein (ELİSA kit) levels

SUMMARY:
There were many studies in the literature discussing the effects of vitamin D deficiency and the role of vitamin D supplementation in SARS-CoV-2 patients. Combined with the possible impact of vitamin D on the pathogenesis of SARS-CoV-2 infection, it is concluded that VDBP-regulated bioavailable and free vitamin D concentrations modulate the human immune system response to viral infections. Because of the gap in the literature, it was emphasized that studies should focus on vitamin D binding protein (VDBP) and gene polymorphism. In this study, it was aimed to investigate the relationship between SARS-CoV-2 infection severity and free and bioavailable vitamin D levels.

DETAILED DESCRIPTION:
It was aimed to investigate the relationship between SARS-CoV-2 infection severity and free and bioavailable vitamin D levels. This study was planned as a case-control study with patients hospitalized in the Haseki Training and Research Hospital Pediatric Infection Service. A total of 82 children, including at least 20 patients in each group were included in the study. The study group was divided into three groups according to COVID-19 WHO clinical progression Scale: unaffected (Group 1), mild (Group 2) and moderate (group 3). In order to investigate the relationship between disease severity and free and bioavailable vitamin D; 25OH vitamin d (μg/L), albumin (g/l) and VDBP levels (ELISA) were used. Vitamin D metabolites were calculated by using Bikle and Vermeulen methods (free Vitamin D BIKLE, free vitamin DVERMEULEN, bioavailable vitamin D). And these three vitamin D parameter levels were compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1-18 years old,
* Positive for SARS-CoV-2 PCR or positive for IgM in the SARS-CoV-2 antibody test (card test or ELISA),
* Do not have a chronic disease (cystic fibrosis, etc.),
* Volunteer to participate in the study.

Exclusion Criteria:

* Being < 1 year of age

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Sars-CoV-2 diagnosed children aged between 1-18 years old and whose parents sign the informed consent form to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
The relationship between free vitamin D levels and SARS CoV-2 infection severity. | baseline (at the time of diagnosis)
  The differences between free vitamin D levels in SARS CoV-2 infected patients according to the symptom severity. SARS CoV-2 infection severity will be categorized according to COVID19 WHO clinical progression Scale as uninfected, mild, moderate to severe.
The relationship between bioavailable vitamin D levels and SARS CoV-2 infection severity. | baseline (at the time of diagnosis)
  The differences between bioavailable vitamin D levels in SARS CoV-2 infected patients according to the symptom severity. SARS CoV-2 infection severity will be categorized according to COVID19 WHO clinical progression Scale as uninfected, mild, moderate to severe.

CONTACTS AND LOCATIONS:
Overall Officials: mahmut caner US, M.D, Principal Investigator — Haseki Education and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Us MC, Devrim Lanpir A, Ozdatli Kurtulus S, Yagci M, Akarsu O, Sahin K, Akkoc G. The role of free vitamin D and vitamin D binding protein in SARS-Cov-2 infection in children. Pediatr Int. 2023 Jan-Dec;65(1):e15680. doi: 10.1111/ped.15680. PMID 37888613
- [Background] May JM. Triacylglycerol turnover in large and small rat adipocytes: effects of lipolytic stimulation, glucose, and insulin. J Lipid Res. 1982 Mar;23(3):428-36. PMID 7042881
- [Background] Alsina M, Martinez-Picado J, Jofre J, Blanch AR. A medium for presumptive identification of Vibrio anguillarum. Appl Environ Microbiol. 1994 May;60(5):1681-3. doi: 10.1128/aem.60.5.1681-1683.1994. PMID 8017947
- [Background] Speeckaert MM, Delanghe JR. Vitamin D binding protein and its polymorphisms may explain the link between vitamin D deficiency and COVID-19. Sci Prog. 2021 Oct;104(4):368504211053510. doi: 10.1177/00368504211053510. No abstract available. PMID 34723751